CLINICAL TRIAL: NCT04859920
Title: Living Conditions of Patients With Diffuse Large B-Cell Lymphoma or Follicular Lymphoma in the Côte d'Or Region
Acronym: LymphoVi
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: MAYNADIE 2020
Record Dates: First submitted 2021-04-22; First posted 2021-04-26 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2022-01

CONDITIONS: Diffuse Large Cell Diffuse Lymphoma; Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular | interventions — Surveys and Questionnaires; Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaires — QLQ-C30, SF-12, HADS, SARASON, EPICES, socio-professional data
Other: Collection of clinical data and treatments — clinical data and treatments

SUMMARY:
The development of new diagnostic tools and targeted therapy have significantly improved the management of non-Hodgkin's malignant lymphomas and thus their long-term prognosis. However, in the study of improved patient management, survival is not the only measurable indicator and preservation of quality of life is an essential component. In addition, there is little existing data regarding the determinants of quality of life in patients with diffuse large B-cell lymphoma (DLBCL) or follicular lymphoma (FL) in the general population in France.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with DLBCL or FL between January 1, 2010 and December 31, 2017,
* Alive as of January 1, 2021,
* Updated patient address.

Exclusion Criteria:

* Other forms of Hematologic Malignancies at diagnosis,
* Minors.
* Person subject to legal protection (curatorship, guardianship)
* Person subject to a judicial safeguard measure
* Pregnant, parturient or breastfeeding woman
* Adults incapable of giving consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Diffuse large cell diffuse B lymphoma Follicular Lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 157 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Generic Questionnaire SF-12 | At inclusion
Specific questionnaire QLQ-C30 | At inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France